CLINICAL TRIAL: NCT04638218
Title: CUHK Jockey Club Tech-based Stroke Rehabilitation Programme - Augmented Reality (AR) Rehabilitation Training System
Brief Title: CUHK Jockey Club Tech-based Stroke Rehabilitation Programme - ARR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019.377
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented Reality (Experimental): The system provides visual and audio feedback which makes the rehabilitation training process more relaxing, interesting and convenient to guide the patients performing appropriate upper-limb, lower-limb exercises and balance training.
  Interventions: Device: Rehabilitation Training System

INTERVENTIONS:
Device: Rehabilitation Training System — The system can capture useful biomechanical data accurately, such as the location of body centre of mass (COM), the body joint angles, and the body posture. These useful data are stored in a database and can be conveniently accessed by the therapists, which facilitate the follow-up of the patients' therapeutic progress.

SUMMARY:
The Hong Kong Jockey Club Charities Trust has supported CUHK to launch a three-year project 'CUHK Jockey Club HOPE4Care Programme' to implement four evidence-based advanced rehabilitation technologies in 40 local elderly day care centres and rehabilitation centres, to benefit the community.

Our research team had developed the "Augmented Reality (AR) Rehabilitation Training System" that can be used as tools for rehabilitation by individuals who have suffered from a stroke or elderly. The system facilitates an active rehabilitative exercise.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of ischemic brain injury or intracerebral haemorrhage shown by magnetic resonance imaging or computed tomography after the onset of stroke;
* Motor impairment in upper-limb, lower-limb, and/or balance;
* No or mild spasticity on the lower-limb or upper-limb (MAS≤2);
* Have sufficient cognition to follow the instructions provided by the rehab system.

Exclusion Criteria

* Any additional medical or psychological condition that would affect their ability to comply with the study protocol, e.g., a significant orthopaedic or chronic pain condition, major post-stroke depression, epilepsy, artificial cardiac pacemaker / joint;
* Severe shoulder or arm contracture/pain;
* Severe knee or hip contracture/pain
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Three months after the last training session
  Berg Balance Scale (BBS), consists of 56-level measures to examine balance ability and to predict falling risk with high reliability (ICC=0.98) (Steffen, Hacker & Mollinger, 2002). Stroke patients were assessed based on their performance on 14 simple mobility tasks, including transfer, standing, and reaching

SECONDARY OUTCOMES:
Modified Ashworth Scale | Three months after the last training session
  Modified Ashworth Scale (MAS), consists of 4-level scale to examine joint spasticity based on muscle tone and resistance detected during passive stretching with good inter-rater reliability (ICC =0.85) (Bohannon & Smith, 1987).
Functional Ambulation Category Test | Three months after the last training session
  Functional Ambulatory Category (FAC) is a reliable measurement of independent walking ability on level-ground walking and stair ambulation, which is a good prediction of independent community walking post-stroke (Mehrholz, et al., 2007). FAC consists of 6-level scale: patients with FAC=4 requires supervision in level ground walking, FAC=5 requires supervision only when walking on non-level surface such as stairs.
Timed 10-meter Walk Test | Three months after the last training session
  Timed 10-Meter Walk Test (10mWT), measures comfortable and fast walking speeds in short distance. The ability to increase walking speed above a comfortable pace suggests the capability to adapt to varying environments, such as crossing street, with high reliability (ICC=0.90-0.96) (Flansbjer, et al., 2005). Average walking speed of healthy elderly subjects ranges in 0.6m/s-1.4m/s, and can increase to 21%-56% above the comfortable pace for faster walking speed
6 Minute Walk Test | Three months after the last training session
  Six-Minute Walk Test (SMWT), measures the maximum walking distance covered in fixed duration as a sub-maximal test of endurance and aerobic capacity. The measurement of 6MWT is highly correlated to FAC (Mehrholz, et al., 2007) with good reliability (ICC=0.94-0.96) (Steffen, Hacker & Mollinger, 2002).
Wolf Motor Function Test (WMFT) | Three months after the last training session
  The WMFT measures upper limb ability through timed and functional tasks. It has 17 items, ranging from 0 to 5 (worse to best).
Action Research Arm Test (ARAT) | Three months after the last training session
  The ARAT has total 19 items, divided into 4 categories (grasp, grip, pinch, and gross arm movement). It ranges from 3 to 0 (best to worse).
Fugl-Meyer Assessment | Three months after the last training session
  Fugl-Meyer Assessment for Upper-Extremity the maximum score is 66, divided into 33 items in the form of a 3-point scale (0-2), 0 is cannot perform and 2 performs fully.
  Fugl-Meyer Assessment for Lower-Extremity consists of 34-level cumulative scoring system to examine lower-limb functions of hemiplegic stroke patients quantitatively through a set of lower-limb movement tasks in reflex, flexor/extensor synergy, volitional movement, coordination and speed (Fugl-Meyer, et al., 1975).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, The Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Derived] Yang ZQ, Du D, Wei XY, Tong RK. Augmented reality for stroke rehabilitation during COVID-19. J Neuroeng Rehabil. 2022 Dec 8;19(1):136. doi: 10.1186/s12984-022-01100-9. PMID 36482468